CLINICAL TRIAL: NCT01137786
Title: A Phase IV Pilot Study to Evaluate Kidney Damage Measured by Neutrophil Gelatinase-Associated Lipocalin (NGAL) as a New Bio-Marker in Patients With Normal eGFR Undergoing Percutaneous Coronary Intervention With IOPAMIDOL Injection 370 or IODIXANOL 320
Brief Title: Kidney Damage in Patients With Normal eGFR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IOP-116
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Stenosis
MeSH Terms: conditions — Coronary Stenosis | interventions — Iopamidol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IOPAMIDOL 370 (Active Comparator)
  Interventions: Drug: Non ionic contrast media comparator
- IODIXANOL 320 (Active Comparator)
  Interventions: Drug: Non ionic contrast media comparator

INTERVENTIONS:
Drug: Non ionic contrast media comparator — One time administration for PCI
  Other Names: Isovue 370
  Arms: IOPAMIDOL 370
Drug: Non ionic contrast media comparator — one time administration for PCI
  Other Names: Visipaque 320
  Arms: IODIXANOL 320

SUMMARY:
This is a pilot study, randomized, double-blind, parallel group comparison of two iodinated contrast agents used during percutaneous coronary intervention (PCI). All patients enrolled must have normal eGFR. Statistical summaries will be presented to analyse the various laboratory tests for the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Provides written Informed Consent and is willing to comply with protocol requirements;
* Is at least 18 years of age;
* Is scheduled to undergo a percutaneous coronary intervention and/or diagnostic coronary angiography.
* Has documented estimated glomerular filtration rate [eGFR] ≥60 mL/min/1.73 m2 calculated with the MDRD formula within 72 hours prior to enrollment.

Exclusion Criteria:

* Is a pregnant or lactating female.
* Has a history of severe congestive heart failure
* Has a history of hyperthyroidism
* Has a history of hypersensitivity to iodinated contrast agents
* Has unstable renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luigia Storto, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Prairie Cardiovascular Consultants, Ltd., Springfield, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Iodixanol 320; Iopamidol 370: Non ionic contrast media comparator : one time administration for PCI
Period: Overall Study
Arm/Group | Iodixanol 320 | Iopamidol 370
Started | 25 | 24
Completed | 24 | 21
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Evaluable patient population for NGAL analysis included all patients with both pre-dose baseline and post-dose blood and/or urine NGAL values for at least 2 out of the 4 planned measurements within 24 hours post-administration.
Groups:
- Iodixanol 320 NGAL Evaluable Population; Iopamidol 370 NGAL Evaluable Population: Non-ionic contrast media comparator: one time administration for PCI
- Total: Total of all reporting groups
Arm/Group | Iodixanol 320 NGAL Evaluable Population | Iopamidol 370 NGAL Evaluable Population | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 10 | 11 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 62.0 (10.65) | 63.4 (12.82) | 62.7 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33
  Italy | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Impact on the Trajectory of Serum and Urinary NGAL Following the Administration of Non-ionic Low Osmolar Contrast Media.
Description: Mean change from baseline values for serum NGAL at 2,4,6,24,48 and 72 hours, and urine NGAL at 2,4,6,24, and 48 hours following the administration of non-ionic low osmolar contrast media.
Time Frame: Baseline and 2, 4, 6, 24, 48, and 72 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Iodixanol 320 Serum NGAL: Serum NGAL (ng/mL) mean change from baseline at 2,4,6,24,48, and 72 hours post-administration of iodixanol 320.
- Iodixanol 320 Urine NGAL: Urine NGAL (ng/mL) mean change from baseline at 2,4,6,24, and 48 hours post-administration of iodixanol 320.
- Iopamidol 370 Serum NGAL: Serum NGAL (ng/mL) mean change from baseline at 2,4,6,24,48, and 72 hours post-administration of iopamidol 370.
- Iopamidol 370 Urine NGAL: Urine NGAL (ng/mL) mean change from baseline at 2,4,6,24, and 48 hours post-administration of iopamidol 370.
Arm/Group | Iodixanol 320 Serum NGAL | Iodixanol 320 Urine NGAL | Iopamidol 370 Serum NGAL | Iopamidol 370 Urine NGAL
Number analyzed (Participants) | 21 | 21 | 21 | 21
ng/mL
  2 hours post-dose | -14.84 (35.46) | -17.71 (49.04) | -9.98 (22.80) | -2.37 (5.45)
  4 hours post-dose | -12.86 (30.57) | -29.33 (64.65) | -5.93 (26.62) | -2.70 (7.09)
  6 hours post-dose | -16.36 (28.77) | -17.90 (51.38) | -5.60 (24.50) | -2.29 (7.66)
  24 hours post-dose | 28.35 (39.21) | -2.10 (46.94) | 20.15 (32.74) | 2.31 (8.70)
  48 hours post-dose | 18.76 (62.77) | -14.60 (34.69) | 34.03 (46.27) | 7.37 (22.84)
  72 hours post-dose | 18.34 (52.28) | NA (NA) — Urine NGAL not measured at this time point as per protocol. | 26.59 (48.13) | NA (NA) — Urine NGAL not measured at this time point as per protocol.

ADVERSE EVENTS:
Arm/Group | Iodixanol 320 | Iopamidol 370
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iodixanol 320 (N=25) | Iopamidol 370 (N=24)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days